CLINICAL TRIAL: NCT02950597
Title: Evaluation of Clinical Impact of Non-Invasive Hemodynamic Monitoring to Optimize Preventative Care of Heart Failure Patients
Brief Title: Clinical Impact of Non-invasive Hemodynamic Monitoring
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Davinder Ramsingh, MD, Study Principal Investigator, Loma Linda University
Other Study IDs: 5160245
Record Dates: First submitted 2016-10-10; First posted 2016-11-01 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Observational Study to Evaluate Utility of Non-invasive Hemodynamic Monitoring

SUMMARY:
Study Details

What is the study design? (eg, randomized, double-blind) Observational Prospective Study

What are the overall objectives of the study? This project is designed to assess the feasibility of using a non-invasive hemodynamic monitoring device in heart failure outpatient clinics. There will be no alteration to patient management for this study. Rather this study seeks to assess the utility of the device by evaluating for the parameters obtained from the device to hospital admission.

How your research will contribute to the advancement of scientific knowledge?

☒This study will confirm/strengthen existing knowledge. ☒This study will test a completely novel hypothesis. ☒This study will explore novel endpoints. ☐Other [please describe]:

DETAILED DESCRIPTION:
B. BACKGROUND:

Nearly five million Americans experience heart failure (HF) and greater than 250,000 die annually. 1 The prevalence has continued to increase with the aging of the US population and HF is now the leading cause of hospitalization among adults >65 in the United states. Despite remarkable improvements in medical therapy, the prognosis of patients with myocardial failure remains poor, with almost 20% of patients dying within 1 year of initial diagnosis and > 80% 8-year mortality. 2 In addition patients who are admitted to the hospital for heart failure have over a 50% readmission rate within six months of discharge. 3,4 These patients require routine clinical care and often require diagnostic and therapeutic procedures. This project seeks to assess if the use of hemodynamic (HD) monitoring technologies (ClearSight/Nexfin) that are currently used in the intraoperative and critical care settings can provide utility by demonstrating associations between alterations in a patients HD values to the likelihood of hospital admission.

The non-invasive HD device utilized (Nexfin, Edwards Lifesciences, Irvine, CA) provided flow-guided cardiovascular parameters that were captured for each clinic visit for up to 24 months. Analysis was performed between the most recent prior clinic visits for patients who were hospitalized for HF exacerbation to those who were not hospitalized. HD data was not used to guide clinical care. A Cox hazard model using a log transformation of HD variables as the covariates, was applied to describe hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in Loma Linda heart failure clinics classified as New York Heart Association (NYHA) Functional Classification of 3 or greater.

Exclusion Criteria:

* Age < 18 years of age,
* pregnancy,
* known severe peripheral artery disease,
* poor perfusion to fingers (as defined as a perfusion index less than 0.5%- www.Masimo.com),
* history of Raynaud's,
* refusal to provide written consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled in the study will include those who are classified as New York Heart Association (NYHA) Functional Classification of three or greater
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-09-19 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
associations between alteration of HD values to hospital admission | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Davinder Ramsingh, MD, Principal Investigator — Loma Linda University Medical Center
Locations (2):
- United States (2):
  - Loma Linda University Department of Anesthesiology, Loma Linda, California
  - Pat Moore, Loma Linda, California

IPD SHARING:
Plan to Share IPD: No